CLINICAL TRIAL: NCT01372514
Title: Institutional Registry of Thromboembolic Disease
Acronym: IRTD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Diego Hernan Giunta, MD, MD, Hospital Italiano de Buenos Aires
Other Study IDs: 995
Record Dates: First submitted 2011-06-10; First posted 2011-06-14 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Thromboembolism; Venous Thromboembolism; Pulmonary Embolism
Keywords: Thromboembolism; Venous Thromboembolism; Pulmonary Embolism
MeSH Terms: conditions — Thromboembolism; Venous Thromboembolism; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- suspected thromboembolic disease: Patients with thromboembolic disease according to diagnostic tests (MDTC with angiography, scintigraphy V/Q, dimer d, ecografia doppler, etc. ) required by the physician.

SUMMARY:
The purpose of this study is to create an institutional registry of Thromboembolic disease through a prospective survey based on epidemiological data, risk factors, diagnosis, prognosis, treatment, monitoring and survival.

The main goal is to describe the occurrence of thromboembolic disease and the characteristics of clinical presentation, evolution and predisposing factors of these episodes in the population of the Hospital Italiano de Buenos Aires.

DETAILED DESCRIPTION:
Deep Vein Thrombosis (DVT) and pulmonary thromboembolism (PTE) are the most common clinical manifestations of thromboembolic disease (TD). The PTE is one of the most important preventable causes of death in hospitalized patients, with a mortality up to 17% in a 3 month period. During the past 20 years important changes have been made in terms of clinical awareness, diagnostic tools and treatment.

No data has been found in our country which shows the TD population incidence. According to WHO, the sex-specific mortality rate associated to TD in Argentina in the year 2001 (including DVT and PE coded by ICD10), estimated by epidemiological death records was 0.2 / 100,000 for men and 0, 5 / 100000 for women (based on 37 and 87 cases respectively). This seems to represent a clear report deficiency.

Registries are systematic surveys which are found in a database. They function as monitoring lists and allow epidemiological evaluations of the affected patients. Several methods can be found to diagnose thromboembolic disease. These include OPTIMEV: Interrogatoire Optimisation de l'évaluation du risque dans l'Maladie ThromboEmbolique of Veineuse (its aim is to include about 10000 cases of suspected DT); MAPPET: Management Strategy and Prognosis of Pulmonary Embolism Registry (its goal is to include 1001 consecutive patients with PE), ICOPER: International Cooperative Pulmonary Embolism Registry (to include 2454 consecutive patients with PE), DVT FREE (including TVP 5451),RIETE: Computerized Patient Record venous thromboembolism in Spain (to register patients with DVT or PE).

No published records have been found regarding the approach used for diagnosis and treatment of suspected PTE patients in our country. Moreover, no publications on systematic epidemiological data (risk factors, assessment and follow-up survival, complications and recurrences)were found.

The registry of suspected TD cases will allow us to distinguish the disease characteristics in our community, the most used diagnostic strategies, the results and the pathology evolution in time.

The Hospital Italiano counts with computerized clinical records which provide incidence, morbidity and mortality data.

It is our belief that this registry will allow us to design studies to improve and standardize the most used diagnostic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Equal to or older than 17 years.
* Followed in HIBA.
* Suspected pulmonary embolism or diagnosed venous thrombosis

Exclusion Criteria:

* Patient with monitoring and care at another facility who only attend the hospital to use its diagnostic method.
* Patient's refusal to participate in the registry or informed consent process.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The eligible population is all patients equal or older than 17 years, evaluated and followed in the Hospital Italiano de Buenos Aires, with an episode of pulmonary embolism suspected by the medical examiner or confirmed diagnosis of DVT or PE. The aim is to include the entire population that meets the criteria for inclusion and no exclusion.
Sampling Method: Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2006-08; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Incidence | 4 years

SECONDARY OUTCOMES:
evaluate new hypothesis | yearly

CONTACTS AND LOCATIONS:
Overall Officials: Diego H Giunta, MD, Principal Investigator — Internal Medicine Clinical research Area Coordinator; Fernan Gonzales Bernaldo de Quirós, MD, Study Director — Internal Medicine Clinical Research Area Chief; Fernando Vazquez, MD, Study Chair — Internal Medicine Staff; Lourdes Posadas-MArtínez, MD, Study Chair — Internal Medicine Clinical research Area , HIBA
Locations (1):
- Hospital Italiano, Buenos Aires, Argentina

REFERENCES:
- [Derived] Grande Ratti MF, Posadas-Martinez ML, Vicens J, Gonzalez Bernaldo de Quiros F, Vazquez FJ, Giunta DH. Incidence of hospital-acquired venous thromboembolic disease. Rev Fac Cien Med Univ Nac Cordoba. 2018 Jun 12;75(2):82-87. doi: 10.31053/1853.0605.v75.n2.17243. PMID 30273531
- [Derived] Vazquez FJ, Posadas-Martinez ML, de Quiros FG, Giunta DH. Prognosis of patients with suspected pulmonary embolism in Buenos Aires: a prospective cohort study. BMC Pulm Med. 2014 Dec 15;14:200. doi: 10.1186/1471-2466-14-200. PMID 25510385
- [Derived] Angriman F, Ferreyro BL, Posadas-Martinez ML, Giunta D, Vazquez FJ, Vollmer WM. Wells Score and Poor Outcomes Among Adult Patients With Subsegmental Pulmonary Embolism: A Cohort Study. Clin Appl Thromb Hemost. 2015 Sep;21(6):539-45. doi: 10.1177/1076029614559772. Epub 2014 Nov 25. PMID 25424529
- [Derived] Ferreyro BL, Angriman F, Giunta D, Posadas-Martinez ML, Vazquez F, De Quiros FG, Amaral AC, Scales DC. Predictive score for estimating cancer after venous thromboembolism: a cohort study. BMC Cancer. 2013 Jul 22;13:352. doi: 10.1186/1471-2407-13-352. PMID 23875619